CLINICAL TRIAL: NCT00358735
Title: Deep Vein Thrombosis (DVT) Prevention in Total Hip Arthroplasty (THA): Continuous Enhanced Circulation Therapy (CECT) Versus Low Molecular Weight Heparin (LMWH)
Brief Title: Deep Vein Thrombosis (DVT) Prevention in Total Hip Arthroplasty: Continuous Enhanced Circulation Therapy (CECT) Versus Low Molecular Weight Heparin (LMWH)
Acronym: SAFE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical Compression Systems (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MedicalCS06CC001
Record Dates: First submitted 2006-07-30; First posted 2006-08-01 (Estimated); Results first posted 2014-10-21 (Estimated); Last update posted 2014-10-30 (Estimated); Status verified 2014-10

CONDITIONS: Deep Vein Thrombosis of Lower Limb; Pulmonary Embolism (PE); Bleeding
Keywords: SAFE; CECT; SFT; ActiveCare; ActiveCare+SFT; Deep Vein Thrombosis prevention; Total Hip Replacement; Total Hip Arthroplasty; Low Molecular Weight Heparin; MCS
MeSH Terms: conditions — Venous Thrombosis; Pulmonary Embolism; Hemorrhage | interventions — Enoxaparin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ActiveCare CECT (Experimental): The ActiveCare CECT device is a mobile compression device used to prevent venous thromboembolic events, used after the induction of anesthesia, throughout the surgery and for 10-12 days after surgery.
  Interventions: Device: ActiveCare CECT device
- LMWH (Enoxaparin) (Active Comparator): Enoxaparin (LMWH) will be used, following a protocol that is considered a standard of care for this patient population. 40mg QD for the remainder of the 10 days.
  Interventions: Drug: Enoxaparin

INTERVENTIONS:
Device: ActiveCare CECT device — Patients will be treated with the ActiveCare+ CECT device starting after the induction of anesthesia, throughout the surgery and for 10-12 days after surgery. Baby aspirin (81 mg) QD can be added (depending on surgeon preference) 12-24 hours after surgery. Post discharge prophylaxis is the same for the remainder of the 10-12 days. Patients will wear the device to the duplex ultrasound when it will be discontinued by nurse.
  Other Names: ActiveCare+; ActiveCare DVT; ActiveCare+SFT
  Arms: ActiveCare CECT
Drug: Enoxaparin — Patients will be treated with Enoxaparin (Lovenox) for a total of 10 days beginning with 30mg BID starting 12-24 hours after surgery and continued until hospital discharge. Post discharge prophylaxis will be Enoxaparin 40mg QD for the remainder of the 10 days.
  Other Names: Lovenox
  Arms: LMWH (Enoxaparin)

SUMMARY:
Evaluation of the safety and effectiveness of ActiveCare+ CECT device +/- baby dose aspirin (81 mg QD) for lowering the potential risk for bleeding and of DVT during and after THA surgery in comparison with LMWH.

DETAILED DESCRIPTION:
Patients undergoing total hip arthroplasty surgery are at particular risk for Thromboembolic disease. To date two prophylactic modalities are being used: mechanical (intermittent pneumatic compression [IPC]) and pharmacological (anticoagulant). Both are effective; however each carries its own advantages and disadvantages.

The purpose of this study is to compare in total hip arthroplasty (THA) patients the safety and effectiveness of the mobile ActiveCare CECT based prophylaxis protocol and compare it with LMWH standard of care protocol for this patient population.

The protocol is based upon the CECT system as the primary DVT prophylaxis method (with or without the addition of low dose baby aspirin [81 mg]).

ELIGIBILITY:
Inclusion Criteria:

Adult patient (Age >18). Patient intended to undergo elective primary unilateral THA surgery. Patient is able and willing to follow instructions of care after surgery. Patient is able and willing to sign the institution human subjects committee approved Informed Consent Form.

Exclusion Criteria:

Patient who has a known coagulation disorder. Patient currently treated with anticoagulant medications. Patient with known thrombophilia Patient with current signs and symptoms of or history of DVT/PE. Patient who is uncooperative or unable to follow instructions. Patient currently suffering from a solid tumor malignancy. Patient with active peptic disease. Patient with known allergy to baby aspirin (81 mg) or enoxaparin. Patient with contraindication to use of the device including patients with leg gangrene, recent skin graft or medical situations where increase venous and lymphatic return is undesirable.Patient has major surgery procedure within 3 months prior to the study surgery, or patients with a major surgery procedure planning during the study period.Pregnant women.Patient who is participating in another clinical drug trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 411 (Actual)
Dates: Start 2006-06; Primary Completion 2008-09 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clifford W Colwell, M.D, Principal Investigator — Scripps Clinic
Locations (9):
- United States (9):
  - Scripps Clinic, La Jolla, California
  - Empire Orthopedic Center, Loma Linda, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - The center for hip and knee surgery, Mooresville, Indiana
  - Center for Joint Preservation and Replacement, Sinai Hospital of Baltimore, Baltimore, Maryland
  - Mayo Clinic, Rochester, Minnesota
  - Hospital for Special Surgery, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - The Center Orthopedic & Neurosurgical Care &Research, Bend, Oregon

REFERENCES:
- [Result] Colwell CW Jr, Froimson MI, Mont MA, Ritter MA, Trousdale RT, Buehler KC, Spitzer A, Donaldson TK, Padgett DE. Thrombosis prevention after total hip arthroplasty: a prospective, randomized trial comparing a mobile compression device with low-molecular-weight heparin. J Bone Joint Surg Am. 2010 Mar;92(3):527-35. doi: 10.2106/JBJS.I.00047. PMID 20194309
- See also: Summary and brochure of the S.A.F.E study — http://www.mcsmed.com/uploadimages/SAFE.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Multi-center study. Recruitment began June 2006 and ended September 2008
Pre-assignment Details: Per protocol:. The pre-randomization evaluation (within 3 days of surgery, may be completed on admission) includes the following:
  * Review of inclusion/exclusion criteria (including evaluation for clinical signs and symptoms of DVT or PE)
  * Demographic parameters
  * Medical history
Groups:
- ActiveCare+SFT (Experimental): The ActiveCare+SFT device is a mobile compression device used to prevent venous thromboembolic events. It was started immediately after the induction of anesthesia, throughout the surgery and for 10-12 days after surgery (in and out hospital).
- LMWH (Enoxaparin) (Active Comparator): Enoxaparin (LMWH) was used, following a protocol that is considered a standard of care for this patient population. 30mg twice a day was given in the hospital and 40mg QD for the remainder of the 10 days (out of hospital).
Period: Overall Study
Arm/Group | ActiveCare+SFT (Experimental) | LMWH (Enoxaparin) (Active Comparator)
Started | 204 | 207
Completed Safety | 198 | 194
Not Completed Safety | 6 | 13
Completed | 196 (Efficacy) | 190 (Efficacy)
Not Completed | 8 | 17

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ActiveCare+SFT (Experimental) | LMWH (Enoxaparin) (Active Comparator) | Total
Number analyzed (Participants) | 198 | 194 | 392
Age, Continuous [Mean (Full Range); unit: years] | 63 [20 to 84] | 62 [32 to 88] | 62.5 [20 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 109 | 105 | 214
  Male | 89 | 89 | 178
body-mass index (Kg/m2) [Mean (Full Range); unit: Kg/m^2] | 28 [17 to 43] | 29 [16 to 49] | 28.5 [16 to 49]
Diagnosis of osteoarthritis (n) [Number; unit: participants]
  Diagnosis | 186 | 184 | 370
  No Diagnosis | 12 | 10 | 22
Duration of surgery (minutes) [Mean (Full Range); unit: Minutes] | 91 [44 to 168] | 96 [41 to 190] | 93.5 [41 to 190]
length of hospital stay (days) [Mean (Full Range); unit: days] | 3.2 [2 to 8] | 3.2 [2 to 10] | 3.2 [2 to 10]

OUTCOME MEASURES:

1. Primary Outcome: Events of Deep Vein Thrombosis (DVT)
Description: 10-12 days post-op: All of the patients underwent Routine bilateral compression Doppler.
  Day of surgery and up to 3 months post-op: Suspected clinical signs and symptoms DVT events were confirmed by standard diagnostic objective methods
Time Frame: 10-12 days post-op; and from day of surgery and up to 3 months if symptomatic
Measure: Number; unit: Events
Units Other Than Participants: Number of Hips Analyzed
Arm/Group | ActiveCare+SFT (Experimental) | LMWH (Enoxaparin) (Active Comparator)
Number analyzed (Participants) | 196 | 190
Number analyzed (Number of Hips Analyzed) | 197 | 192
Events
  Total DVT | 8 | 8
  Distal DVT | 5 | 6
  Proximal DVT | 3 | 2
Statistical Analysis 1: Comparison: ActiveCare+SFT (Experimental) vs LMWH (Enoxaparin) (Active Comparator); Test type: Superiority or Other; p > 0.05, Chi-squared

2. Primary Outcome: Clinical PE (Pulmonary Embolism) Events
Description: Clinical PE events PE (Pulmonary Embolism) events were confirmed by spiral CT
Time Frame: Day of surgery and up to 3 months
Measure: Number; unit: Events
Units Other Than Participants: Number of Hips Analyzed
Arm/Group | ActiveCare+SFT (Experimental) | LMWH (Enoxaparin) (Active Comparator)
Number analyzed (Participants) | 196 | 190
Number analyzed (Number of Hips Analyzed) | 197 | 192
Events | 2 | 2
Statistical Analysis 1: Comparison: ActiveCare+SFT (Experimental) vs LMWH (Enoxaparin) (Active Comparator); Test type: Superiority or Other; p > 0.05, Chi-squared

3. Secondary Outcome: Major Bleeding Complication
Description: Major bleeding is defined as bleeding that requires rehospitalization or prolonged hospitalization, requires any intervention such as surgery or hematoma aspiration to prevent permanent impairment or damage, endangered critical organs, is life threatening or causes death. Data collected included bleeding index, a decrease in hemoglobin greater than/equal to 20 g/L, and number of units of blood transfused.
Time Frame: Up to 30 days
Measure: Number; unit: Events
Units Other Than Participants: Number of Hips Analyzed
Arm/Group | ActiveCare+SFT (Experimental) | LMWH (Enoxaparin) (Active Comparator)
Number analyzed (Participants) | 198 | 194
Number analyzed (Number of Hips Analyzed) | 199 | 196
Events | 0 | 11
Statistical Analysis 1: Comparison: ActiveCare+SFT (Experimental) vs LMWH (Enoxaparin) (Active Comparator); Test type: Superiority or Other; p = 0.0004, Chi-squared

4. Secondary Outcome: OutPatient Patients' Compliance
Description: Total usage time with the pneumatic device (patient's compliance) was recorded using the ActiveCare+SFT device internal timer.
  The compliance was calculate as total actual operation time (for the entire arm/group) divided by the total time passes since the initiation of home treatment (for the entire arm/group).
  The compliance is expressed as percentages.
Time Frame: 10-12 days post-op
Measure: Number; unit: percentage of usage time
Arm/Group | ActiveCare+SFT (Experimental)
Number analyzed (Participants) | 180
percentage of usage time | 83

5. Post Hoc Outcome: Events of Clinical Sign and Symptoms of VTE (DVT and/or PE)
Description: Events of clinical Sign and symptoms of VTE (DVT and/or PE), confirmed by standard objective diagnostic methods
Time Frame: Day of surgery and up to 3 months
Measure: Number; unit: Events
Units Other Than Participants: Number of Hips Analyzed
Arm/Group | ActiveCare+SFT (Experimental) | LMWH (Enoxaparin) (Active Comparator)
Number analyzed (Participants) | 199 | 196
Number analyzed (Number of Hips Analyzed) | 197 | 192
Events | 10 | 10
Statistical Analysis 1: Comparison: ActiveCare+SFT (Experimental) vs LMWH (Enoxaparin) (Active Comparator); Test type: Superiority or Other; p = 0.953, Chi-squared

6. Post Hoc Outcome: Total Number of Blood Transfusion Units
Description: Number of blood units used (Autologous units and allogeneic units) (blood units during surgery not included)
Time Frame: Between the immediate postoperative measurement and discharge
Measure: Number; unit: Units
Units Other Than Participants: Number of Hips Analyzed
Arm/Group | ActiveCare+SFT (Experimental) | LMWH (Enoxaparin) (Active Comparator)
Number analyzed (Participants) | 198 | 194
Number analyzed (Number of Hips Analyzed) | 199 | 196
Units | 82 | 122
Statistical Analysis 1: Comparison: ActiveCare+SFT (Experimental) vs LMWH (Enoxaparin) (Active Comparator); Test type: Superiority or Other; p = 0.050, Chi-squared

7. Post Hoc Outcome: Allogeneic Blood Transfusion Units
Description: Allogeneic blood transfusion per patient in specific treatment Group
Time Frame: Up to 30 days
Measure: Mean (Standard Deviation); unit: Avg. Unit per patient in arm
Arm/Group | ActiveCare+SFT (Experimental) | LMWH (Enoxaparin) (Active Comparator)
Number analyzed (Participants) | 198 | 194
Avg. Unit per patient in arm | 0.13 (0.48) | 0.32 (0.8)
Statistical Analysis 1: Comparison: ActiveCare+SFT (Experimental) vs LMWH (Enoxaparin) (Active Comparator); Test type: Superiority or Other; p = 0.010, Chi-squared

8. Post Hoc Outcome: Autologous Blood Transfusion Units
Description: Autologous blood transfusion per patient in specific treatment Group
Time Frame: Up to 30 days
Measure: Mean (Standard Deviation); unit: Avg. Unit per patient in arm
Arm/Group | ActiveCare+SFT (Experimental) | LMWH (Enoxaparin) (Active Comparator)
Number analyzed (Participants) | 198 | 194
Avg. Unit per patient in arm | 0.28 (0.53) | 0.3 (0.52)
Statistical Analysis 1: Comparison: ActiveCare+SFT (Experimental) vs LMWH (Enoxaparin) (Active Comparator); Test type: Superiority or Other; p = 0.507, Chi-squared

9. Post Hoc Outcome: Bleeding Index ≥ 2
Description: Bleeding index was defined as the number of units of whole blood or packed red blood cells transfused plus the difference between the first hemoglobin value after surgery and the value prior to discharge
Time Frame: Surgery till discharge
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ActiveCare+SFT (Experimental) | LMWH (Enoxaparin) (Active Comparator)
Number analyzed (Participants) | 198 | 194
units on a scale | 1.3 (1.04) | 1.5 (1.27)
Statistical Analysis 1: Comparison: ActiveCare+SFT (Experimental) vs LMWH (Enoxaparin) (Active Comparator); Test type: Superiority or Other; p = 0.052, Chi-squared

10. Post Hoc Outcome: Changes in Hemoglobin Levels
Description: Changes in Hemoglobin levels
Time Frame: After surgery untill discharge
Measure: Mean (Standard Deviation); unit: mean change (g/l)
Arm/Group | ActiveCare+SFT (Experimental) | LMWH (Enoxaparin) (Active Comparator)
Number analyzed (Participants) | 198 | 194
mean change (g/l) | 8 (1.26) | 9 (1.47)
Statistical Analysis 1: Comparison: ActiveCare+SFT (Experimental) vs LMWH (Enoxaparin) (Active Comparator); Test type: Superiority or Other; p = 0.798, Chi-squared

11. Post Hoc Outcome: Composite Outcome of Major Bleeding + VTE
Description: Major bleeding + DVT events + PE Events
Time Frame: Day of surgery and up to 3 months
Measure: Number; unit: Events
Arm/Group | ActiveCare+SFT (Experimental) | LMWH (Enoxaparin) (Active Comparator)
Number analyzed (Participants) | 196 | 190
Events | 10 | 21
Statistical Analysis 1: Comparison: ActiveCare+SFT (Experimental) vs LMWH (Enoxaparin) (Active Comparator); Test type: Superiority or Other; p = 0.036, Chi-squared

12. Secondary Outcome: Serious Adverse Events
Description: Serious Adverse Events (SAE) is any event that prolongs hospitalization or requires re-hospitalization, that requires intervention to prevent permanent impairment or damage, that causes permanent disability, or that is life threatening.
  SAE did not include Venous thrombolembolism (VTE) events (DVT and PE) and Major bleeding complications as these are outcome measures
Time Frame: SAE data were collected Up to 3 months post-op
Measure: Number; unit: events
Arm/Group | ActiveCare+SFT (Experimental) | LMWH (Enoxaparin) (Active Comparator)
Number analyzed (Participants) | 198 | 194
events | 3 | 10

13. Secondary Outcome: In-Patients' Compliance
Description: Total usage time with the pneumatic device (patient's compliance) was recorded using the ActiveCare+SFT device internal timer.
  The compliance was calculate as total actual operation time (for the entire arm/group) divided by the total time passes since the initiation of treatment at hospital (for the entire arm/group).
  The compliance is expressed as percentages.
Time Frame: Surgery till discharge
Measure: Number; unit: percentage of usage time
Arm/Group | ActiveCare+SFT (Experimental)
Number analyzed (Participants) | 180
percentage of usage time | 91

ADVERSE EVENTS:
Time Frame: SAE data were collected Up to 3 months post-op
Description: SAE did not include VTE events(DVT and PE) and Major bleeding complications as these are outcome measures
Arm/Group | ActiveCare+SFT (Experimental) | LMWH (Enoxaparin) (Active Comparator)
Serious Adverse Events (participants affected / at risk) | 3/198 | 10/194
Other Adverse Events (participants affected / at risk) | 89/198 | 102/194
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ActiveCare+SFT (Experimental) (N=198) | LMWH (Enoxaparin) (Active Comparator) (N=194)
Cardiac Disorders (Cardiac disorders) | 0 | 1
Dislocation (Musculoskeletal and connective tissue disorders) | 0 | 5
Fever due to aspiration (Infections and infestations) | 1 | 0
Parkinson (new event) (Nervous system disorders) | 1 | 0
Stress fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
supraventricular cardiac arrhythmia (Cardiac disorders) | 1 | 2
Thrombocytopenia (HIT?) (Blood and lymphatic system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ActiveCare+SFT (Experimental) (N=198) | LMWH (Enoxaparin) (Active Comparator) (N=194)
Minor Bleeding (Blood and lymphatic system disorders) | 74 (74) | 78 (78) — Minor bleeding was any bleeding that was not major bleeding (e.g., increased wound drainage reported by the surgeon or a drop in the hemoglobin level not requiring transfusion or prolonged hospitalization).
Edema (Blood and lymphatic system disorders) | 7 (7) | 22 (22)
Skin irritation (Skin and subcutaneous tissue disorders) | 8 (8) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No